CLINICAL TRIAL: NCT03231540
Title: Effect of Whey Protein-enriched Enteral Nutrition in Addition to Standardized Exercise Training on the PREServation of MUScle Function in Critically Ill Patients: A Randomized Controlled Trial
Brief Title: The PREServation of MUScle Function in Critically Ill Patients (PRESMUS)
Acronym: PRESMUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Sandra Stapel, intensivist, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016.101
Record Dates: First submitted 2017-04-21; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Critically Ill
Keywords: Critical care; nutrition; whey protein; mechanical ventilation; muscle function
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): whey protein supplement enriched enteral nutrition, with protein intake of 1.5g/kg/day; in addition to standardized exercise training
  Interventions: Dietary Supplement: Whey protein supplement
- control group (No Intervention): standard enteral nutrition, with protein intake of 1g/kg/day; in addition to standardized exercise training

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — Whey protein supplement to target protein intake of 1.5 g/kg/day
  Other Names: Beneprotein Nestle
  Arms: intervention group

SUMMARY:
This study evaluates the effect of whey protein enriched enteral nutrition in addition to exercise training on the preservation of muscle function in critically ill patients.

One half of patients receive whey protein enriched enteral nutrition with a protein intake of 1.5 g/kg/day and the other half of patients receive standard enteral nutrition with a protein intake of 1 g/kg/day.

DETAILED DESCRIPTION:
Muscle wasting has an enormous impact on long-term physical performance and quality of life of intensive care survivors. Limitation of muscle wasting might therefore improve physical performance and quality of life. Data on high protein nutritional intake in addition to a standardized exercise training program to prevent skeletal muscle wasting during critical illness are lacking.

Objective: to determine whether early high protein intake, using an enteral whey protein supplement, in addition to a standardized exercise training program and standard enteral nutrition preserves: a) in vitro skeletal muscle function in critically ill patients during the first week of intensive care unit (ICU) admission and b) short- and long-term in vivo muscle function and mass, clinical outcomes and quality of life in critically ill patients. Secondly, to determine whether high protein intake, in addition to standardized exercise and standard enteral nutrition, increases muscle protein synthesis and attenuates activation of the Ubiquitin-Proteasome pathway in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the intensive care
* Mechanically ventilated
* Expected duration of ventilation of 72 hours
* Expected to tolerate and require enteral nutrition for more than 72 hours
* Sequential organ failure assessment (SOFA)-score>6 on admission day
* Written informed consent of patient or legal representative

Exclusion Criteria:

* Contra-indication to enteral nutrition
* Short bowel syndrome
* Child C liver cirrhosis or acute liver failure
* Dialysis dependency
* Requiring other specific enteral nutrition for medical reason
* Body mass index (BMI) > 35 kg/m2
* Extensive treatment limitations
* Disseminated malignancy
* Haematological malignancy
* Primary neuromuscular pathology
* Chronic use of corticosteroids for > 7 days before ICU admission
* Contra-indication for muscle biopsy (need for uninterrupted systemic anticoagulation, prothrombin time >1.4 , Thrombocytes <100).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
in vitro loss of skeletal muscle function | day 1-3 and day 8-10
  measured by contractility of of individual muscle fibers

SECONDARY OUTCOMES:
loss of muscle function | day 1-3, day 8-10, day 28
  Medical research council (MRC) sum score,
changes in body composition | day 1-3, day 8-10, day 28
  Bioelectrical impedance analysis (BIA)
loss of muscle mass | day 1-3, day 8-10, day 28
  Ultrasound (US) of the quadriceps femoris muscle and diaphragm, questionnaires
quality of life | 3 months
  Short form (SF)- 36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sandra N Stapel, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided